CLINICAL TRIAL: NCT03533777
Title: Comparison of Retrograde and Antegrade Peripheral Intravenous Cannulation on the Ability to Aspirate Blood Samples in the Operating Room
Brief Title: Antegrade Versus Retrograde IV for Blood Draws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Andrew Feider, assistant professor of anesthesia, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201805706
Record Dates: First submitted 2018-04-25; First posted 2018-05-23 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: There is no Focus on Any Specific Condition
MeSH Terms: interventions — Blood Specimen Collection; Saline Solution

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either antegrade or retrograde IV catheter placement. Although 267 patients were consented/enrolled in the study, only 230 patients were ultimately randomized. 37 patients were withdrawn from the study prior to randomization because they no longer met inclusion/exclusion criteria.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Placement of the IV catheter will occur after the subject is placed under general anesthesia and will be removed immediately upon arrival in the post-anesthesia care unit (PACU). Thus, the study participant will be unaware of which study arm they were in. An anesthesiologist member of the research team will place the IV immediately after randomization in the operating room. They will have a drape obscuring the view from the clinical anesthesia provider and will cover the IV with an opaque towel after insertion. Thus, the care provider will not have knowledge of which treatment arm their patient is randomized to. Intraoperative data will be gathered by the anesthesia care provider and postoperative questionnaire data will be gathered by a research coordinator member of the study team. The anesthesiologist who placed the study IV will not gather or have access to any of the subsequent data gathered on the study subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antegrade Intravenous Catheter (Active Comparator): A 20 gauge 30 millimeter peripheral intravenous catheter will be placed in an upper extremity vein in standard antegrade fashion (with the tip pointed towards the direction of blood flow). Blood draws from this IV catheter will be attempted twice throughout the study. An infusion of 0.9% normal saline will be connected to the catheter and infused at a rate of 20 milliliters per hour to keep open (TKO) for future use by preventing blood clot development within the catheter.
  Interventions: Procedure: Peripheral intravenous catheter placement; Other: Blood draw; Device: Peripheral intravenous catheter; Drug: To keep open (TKO) infusion of 0.9% normal saline
- Retrograde Intravenous Catheter (Experimental): A 20 gauge 30 millimeter peripheral intravenous catheter will be placed in an upper extremity vein in a retrograde fashion (with the tip pointed away from the direction of blood flow). Blood draws from this IV catheter will be attempted twice throughout the study. An infusion of 0.9% normal saline will be connected to the catheter and infused at a rate of 20 milliliters per hour to keep open (TKO) for future use by preventing blood clot development within the catheter.
  Interventions: Procedure: Peripheral intravenous catheter placement; Other: Blood draw; Device: Peripheral intravenous catheter; Drug: To keep open (TKO) infusion of 0.9% normal saline

INTERVENTIONS:
Procedure: Peripheral intravenous catheter placement — The region of the upper extremity in which the IV will be placed will be prepped with chlorhexidine and a proximal elastic tourniquet is applied to the upper arm. A 20 gauge 30 millimeter IV catheter is inserted into an upper extremity vein by an anesthesiologist in either an antegrade or retrograde direction depending on which treatment arm the study subject is randomized to.
Other: Blood draw — A 20 milliliter(mL) syringe will be connected to the study IV tubing and used to aspirate 20 mL of blood from the study IV catheter. If 20 mL are unable to be aspirated over a 2 minute time frame, a proximal rubber tourniquet will be applied to the upper arm and the blood draw will be reattempted.This will occur twice throughout the study.
Device: Peripheral intravenous catheter — A 20 gauge 30 millimeter long BD Insyte(TM) Autoguard(TM) angiocatheter will be used for peripheral intravenous catheter placement as described above.
Drug: To keep open (TKO) infusion of 0.9% normal saline — After placement of the peripheral intravenous catheter, an infusion of 0.9% normal saline will be connected to the catheter and infused at a rate of 20 milliliters per hour to keep open (TKO) for future use by preventing blood clot development within the catheter.

SUMMARY:
The purpose of this study is to compare success rates of antegrade and retrograde intravenous (IV) catheters in their ability to aspirate 20 milliliter blood sample within a 2 minute time frame, 3 hours after initial insertion. Antegrade IV catheters are placed identically to conventional IV catheters, with the end of the catheter pointed toward the direction of blood flow to the heart. Retrograde catheters are placed "backwards" with the end of the catheter pointed away from the direction of venous blood flow. The hypothesis is that retrograde IVs will have a significantly higher success rate of blood draw at the 3 hour time mark without use of a proximal tourniquet.

DETAILED DESCRIPTION:
1. Patients scheduled for surgery under general anesthesia at the University of Iowa Hospitals and Clinics (UIHC) will be recruited pre-operatively in the Day of Surgery Admissions (DoSA) rooms before their surgery takes place. Once the subject is recruited and has signed a consent form, they will be randomized to either retrograde or antegrade IV. Once in the operating room and general anesthesia has been induced, a 20 gauge 30 millimeter catheter will be placed in a vein of one of the upper extremities by an anesthesiologist member of the research team. A drape will obscure viewing of the procedure by the clinical anesthesia provider. They will then connect the catheter to an IV tubing set and cover the insertion site with a opaque towel, so as to blind the anesthesia provider caring for the patient in the OR.
2. 0.9% normal saline (NS) will be infused at a rate of 20 milliliters (mL) per hour to keep it open (TKO) and it will not be used for drug infusion.
3. Three hours after insertion, the anesthesia provider in the OR will attempt a blood draw from a stopcock 33 inches from the catheter. A successful 20 mL blood draw must be achieved within 2 minutes after attempt is started or it will be defined as a failed attempt. If blood draw fails, an upper arm tourniquet will be placed and the blood draw will be reattempted following the same guidelines as the initial attempt. After every blood draw, 10 mL of NS will be flushed back through the IV.
4. At the end of surgery, within 30 minutes of extubation, the anesthesia provider in the OR will attempt a blood draw from a stopcock 33 inches from the catheter. A successful 20 mL blood draw must be achieved within 2 minutes after attempt is started or it will be defined as a failed attempt. If blood draw fails, an upper arm tourniquet will be placed and the blood draw will be reattempted following the same guidelines as the initial attempt. After every successful blood draw 10 mL of NS will be flushed back through the IV.
5. The IV will be saline locked at the end of the case.
6. The IV will be removed within 15 minutes upon arrival in the Post Anesthesia Care Unit (PACU) by the same anesthesiologist member of the research team who placed it and the site will be dressed appropriately.
7. Follow up will happen on post-operative Day 1 (POD1) either in person if the patient is admitted to a UIHC inpatient unit or via a phone call if they are discharged before POD1. At this POD1 check, the patient will be asked about the prior IV site: level of pain, if there is a hematoma, or possible infection. There will be a maximum of 3 attempts to contact the subject. This data will be gathered by a research coordinator member of the research team who is unaware of which study arm the subject was randomized to.
8. A second follow up will happen on 14 days after the surgery/IV placement via a phone call. Again, the patient will be asked about the prior IV site: level of pain, if there is a hematoma, or possible infection. There will be a maximum of 3 attempts to contact the subject. This data will be gathered by a research coordinator member of the research team who is unaware of which study arm the subject was randomized to.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* English speaking
* Age 18-90
* Scheduled to undergo surgery under general anesthesia at the University of Iowa Hospitals and Clinics
* Surgery is scheduled to last at least 3 hours

Exclusion Criteria:

* Emergency surgery
* Previous or planned sentinel node dissection on ipsilateral arm of study IV
* Existing or planned arteriovenous fistula on ipsilateral arm of study IV
* Surgery with lateral positioning
* Surgery which involves tucking the arm with study IV
* Any additional peripheral IV catheters distal to study IV
* Non invasive blood pressure cuff placed on arm with study IV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Ability to aspirate blood samples without tourniquet 3 hours after IV insertion | three hours after IV insertion
  As compared to IV catheters placed in the standard antegrade fashion, do IV catheters placed in a retrograde direction have a higher blood draw success rate 3 hours after initial insertion, without the use of a tourniquet? Investigators define "blood draw success" as the ability to aspirate 20 mL blood samples within a 2 minute time frame. It is defined as a binary outcome variable: success vs failure. For the primary comparison of success rates in the retrograde vs antegrade IV groups, chi-square test will be used.

SECONDARY OUTCOMES:
Ability to aspirate blood samples without tourniquet at the end of surgery | three to eight hours after IV insertion
  As compared to IV catheters placed in the standard antegrade fashion, do IV catheters placed in a retrograde direction have a higher blood draw success rate greater than 3 hours after initial insertion, without the use of a tourniquet? Investigators define "blood draw success" as the ability to aspirate 20 mL blood samples within a 2 minute time frame. It is defined as a binary outcome variable: success vs failure. For the primary comparison of success rates in the retrograde vs antegrade IV groups, chi-square test will be used.
Ability to aspirate blood samples with tourniquet (if needed) 3 hours after IV insertion | three hours after IV insertion
  As compared to IV catheters placed in the standard antegrade fashion, do IV catheters placed in a retrograde direction have a higher blood draw success rate 3 hours after initial insertion, with the use of a tourniquet (if needed)? Investigators define "blood draw success" as the ability to aspirate 20 mL blood samples within a 2 minute time frame. It is defined as a binary outcome variable: success vs failure. For the primary comparison of success rates in the retrograde vs antegrade IV groups, chi-square test will be used.
Ability to aspirate blood samples with tourniquet (if needed) at the end of surgery | three to eight hours after IV insertion
  As compared to IV catheters placed in the standard antegrade fashion, do IV catheters placed in a retrograde direction have a higher blood draw success rate greater than 3 hours after initial insertion, with the use of a tourniquet (if needed)? Investigators define "blood draw success" as the ability to aspirate 20 mL blood samples within a 2 minute time frame. It is defined as a binary outcome variable: success vs failure. For the primary comparison of success rates in the retrograde vs antegrade IV groups, chi-square test will be used.
Body mass index (BMI) as a predictor of success rate of blood draws 3 hours after IV insertion. | three hours after IV insertion
  As an exploratory analyses, the effect of BMI as a predictor of success rate of blood draws will be assessed by including the BMI in the logistic regression model where the outcome of interest is the successful blood draw 3 hours after initial insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feider, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelaal Ahmed Mahmoud A, El-Shafei HI, Yassin HM, Elramely MA, Abdelhaq MM, El Kady HW, Awada WNF. Comparison Between Retrograde and Antegrade Peripheral Venous Cannulation in Intensive Care Unit Patients: Assessment of Thrombus Formation. Anesth Analg. 2017 Jun;124(6):1839-1845. doi: 10.1213/ANE.0000000000001703. PMID 27941574
- [Background] Nauck MA, Liess H, Siegel EG, Niedmann PD, Creutzfeldt W. Critical evaluation of the 'heated-hand-technique' for obtaining 'arterialized' venous blood: incomplete arterialization and alterations in glucagon responses. Clin Physiol. 1992 Sep;12(5):537-52. doi: 10.1111/j.1475-097x.1992.tb00357.x. PMID 1395446
- [Background] Brooks DC, Black PR, Arcangeli MA, Aoki TT, Wilmore DW. The heated dorsal hand vein: an alternative arterial sampling site. JPEN J Parenter Enteral Nutr. 1989 Jan-Feb;13(1):102-5. doi: 10.1177/0148607189013001102. PMID 2926973
- [Background] Liu D, Moberg E, Kollind M, Lins PE, Adamson U, Macdonald IA. Arterial, arterialized venous, venous and capillary blood glucose measurements in normal man during hyperinsulinaemic euglycaemia and hypoglycaemia. Diabetologia. 1992 Mar;35(3):287-90. doi: 10.1007/BF00400932. PMID 1563586
- [Background] Copeland KC, Kenney FA, Nair KS. Heated dorsal hand vein sampling for metabolic studies: a reappraisal. Am J Physiol. 1992 Nov;263(5):E1010-4. doi: 10.1152/ajpendo.1992.263.5.E1010. PMID 1443110
- [Background] Diamond MP, Kruger M, Collins K, Brossoit M, Subramanian M. Antecubital vein venous sampling does not distort circulating levels of peptide and sex steroid hormones. Fertil Steril. 2005 May;83(5):1557-60. doi: 10.1016/j.fertnstert.2005.01.001. PMID 15866606
- [Background] Abumrad NN, Rabin D, Diamond MP, Lacy WW. Use of a heated superficial hand vein as an alternative site for the measurement of amino acid concentrations and for the study of glucose and alanine kinetics in man. Metabolism. 1981 Sep;30(9):936-40. doi: 10.1016/0026-0495(81)90074-3. No abstract available. PMID 7022111
- [Background] Nuttall G, Burckhardt J, Hadley A, Kane S, Kor D, Marienau MS, Schroeder DR, Handlogten K, Wilson G, Oliver WC. Surgical and Patient Risk Factors for Severe Arterial Line Complications in Adults. Anesthesiology. 2016 Mar;124(3):590-7. doi: 10.1097/ALN.0000000000000967. PMID 26640979
- [Background] Bhananker SM, Liau DW, Kooner PK, Posner KL, Caplan RA, Domino KB. Liability related to peripheral venous and arterial catheterization: a closed claims analysis. Anesth Analg. 2009 Jul;109(1):124-9. doi: 10.1213/ane.0b013e31818f87c8. Epub 2009 Apr 17. PMID 19377051
- [Background] Abolfotouh MA, Salam M, Bani-Mustafa A, White D, Balkhy HH. Prospective study of incidence and predictors of peripheral intravenous catheter-induced complications. Ther Clin Risk Manag. 2014 Dec 8;10:993-1001. doi: 10.2147/TCRM.S74685. eCollection 2014. PMID 25525365
- [Background] Raffa m, Greco M, Barbati A. Intravenous Retrograde Anesthesia. In: Alemanno F, Bosco M, Barbati A, eds. Anesthesia of the Upper Limb. Verlag, Italia: Springer; 2014 225-230.
- See also: Understanding retrograde I.V. blood collection in clinical research. — https://www.americannursetoday.com/understanding-retrograde-v-blood-collection-clinical-research/.